CLINICAL TRIAL: NCT02625558
Title: A Double Blind, Placebo Controlled Trial of Oral Riociguat for Sarcoidosis Associated Pulmonary Hypertension
Brief Title: Riociguat for Sarcoidosis Associated Pulmonary Hypertension
Acronym: RioSAPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-7130
Record Dates: First submitted 2015-05-26; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis
Keywords: riociguat; saph; sarcoidosis; sarcoidosis associated pulmonary hypertension
MeSH Terms: conditions — Sarcoidosis | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riociguat (Active Comparator): Active drug
  Interventions: Drug: Riociguat
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat — Patients will initiated on 0.5 mg tid and titrated every 2 weeks to a maximum of 2.5 mg three times a day
  Other Names: Rio
  Arms: Riociguat
Drug: Placebo — Placebo given three times a day
  Arms: Placebo

SUMMARY:
Double blind placebo controlled trial of riociguat for sarcoidosis associated pulmonary hypertension

DETAILED DESCRIPTION:
Study design Patients will be recruited into double blind randomized trial of riociguat with 1:1 active drug to placebo. The table below summarizes the study design. Patients will have previously undergone right heart catheterization (RHC) within six months of initial dose dispensation and with no significant change in treatment for pulmonary hypertension. Patients will initiated on 0.5 mg tid and titrated every 2 weeks to a maximum of 2.5 mg three times a day.

The patient will be treated for 48 weeks or until clinical worsening of disease. An adjudication committee will review all cases of clinical worsening. This committee will be blinded to treatment. The determination by the adjudication committee will be used as the final determinant for the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of sarcoidosis
* Age ≥ 18 years.
* Life expectancy of at least 2 years.
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Females of reproductive potential (FRP) must have a negative, pre-treatment pregnancy test.
* FRP must obtain monthly pregnancy tests during treatment and one month after treatment discontinuation. Post-menopausal women (defined as no menses for at least 1 year or post-surgical from bilateral oophorectomy) and surgically sterilized women are not required to undergo a pregnancy test.
* Females of reproductive potential and all non-vasectomized male participants must agree to use reliable contraception when sexually active.
* Subjects (males and females) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 30 days after the last dose of study drug.
* Willing and able to comply with the protocol, including follow-up visits and examinations

Exclusion Criteria:

* Patients with an FVC of less than 30% of predicted during screening visit.
* Patients with severe airway obstruction
* Patients unable to perform the 6 minute walk test
* Pregnant women (i.e. positive serum ß-human chorionic gonadotropin test or other signs of pregnancy),
* Breast feeding women
* FRP not using reliable contraception as recommended in the Prescriber Guide for the riociguat pregnancy monitoring program
* Subjects with a medical disorder, condition, or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator
* Known significant left heart disease:
* Pulmonary venous hypertension indicated by baseline pulmonary capillary wedge pressure > 15 mmHg
* Active state or history of hemoptysis or pulmonary hemorrhage
* Subjects requiring nitrates for any reason
* Subject using nitrates within one month of entering study
* Pulmonary veno-occlusive disease
* Subjects with underlying medical disorders with an anticipated life expectancy below 2 years (e.g. active cancer disease with localized and/or metastasized tumor).
* Subjects with hypersensitivity to the investigational drug or any of the excipients.
* Women who are pregnant or breast-feeding.
* Severe proven or suspected coronary artery disease
* Clinical relevant hepatic dysfunction indicated by: bilirubin >2 times upper limit normal at Visit 0 and/or: alanine aminotransferase (ALT) or AST aspartate aminotransferase (AST) >3 times upper limit normal at Visit 0 and/or: signs of severe hepatic insufficiency (e.g. impaired albumin synthesis with an albumin <32 g/L, hepatic encephalopathy > grade 1a) at Visit 0

West Haven Criteria of Altered Mental Status in Hepatic Encephalopathy

* Severe renal insufficiency indicated by a glomerular filtration rate <30 mL/min at Visit 0, e.g. calculated based on the Cockcroft formula or the Modification of Diet in Renal Disease Study Group (MDRD) formula
* Inability to comply with the protocol and/or not willing or not available for follow-up assessments.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.

Excluded therapies and medications, previous and concomitant

* Specific (e.g. sildenafil or tadalafil) or unspecific phosphodiesterase inhibitors (e.g. dipyridamole, theophylline).
* NO donors (e.g. nitrates). Single applications of vasoactive drugs in connection with diagnostic vasoreactive testing are allowed.
* Concurrent use of another investigational drug or device therapy (i.e., outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).
* Major surgery within 30 days prior to start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Time until clinical worsening | 48 weeks
  Patient shows deterioration using fixed criteria

SECONDARY OUTCOMES:
Safety: adverse events | 48 weeks
  adverse events
Pulmonary function | 48 weeks
  Changes in FVC
Quality of life | 48 weeks
  Changes in QOL using general and sarcoidosis specific instruments
Six minute walk | 48 weeks
  Change in six minute walk distance

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — University of Cincinnati; Steve Nathan, MD, Principal Investigator — Inova Fairfax Hospital
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Baughman RP, Shlobin OA, Gupta R, Engel PJ, Stewart JI, Lower EE, Rahaghi FF, Zeigler J, Nathan SD. Riociguat for Sarcoidosis-Associated Pulmonary Hypertension: Results of a 1-Year Double-Blind, Placebo-Controlled Trial. Chest. 2022 Feb;161(2):448-457. doi: 10.1016/j.chest.2021.07.2162. Epub 2021 Aug 4. PMID 34363816